CLINICAL TRIAL: NCT02623699
Title: A Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB067 Administered to Adult Subjects With Amyotrophic Lateral Sclerosis and Confirmed Superoxide Dismutase 1 Mutation
Brief Title: An Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of BIIB067 (Tofersen) in Adults With Inherited Amyotrophic Lateral Sclerosis (ALS)
Acronym: VALOR (Part C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 233AS101; 2015-004098-33 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2015-12-08 (Estimated); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: IONIS-SOD1Rx; SOD1; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tofersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part A-SAD: Combined Placebo (Placebo Comparator): Participants will be administered tofersen-matching placebo once by intrathecal bolus injection on Day 1 of Cohorts 1, 2, 3, and 4 respectively.
  Interventions: Drug: Placebo
- Part A-SAD: Cohort 1: Tofersen 10 mg (Experimental): Participants will be administered tofersen 10 mg once by intrathecal bolus injection on Day 1.
  Interventions: Drug: Tofersen
- Part A-SAD: Cohort 2: Tofersen 20 mg (Experimental): Participants will be administered tofersen 20 mg once by intrathecal bolus injection on Day 1 of Cohort 2 after the safety review of Cohort 1.
  Interventions: Drug: Tofersen
- Part A-SAD: Cohort 3: Tofersen 40 mg (Experimental): Participants will be administered tofersen 40 mg once by intrathecal bolus injection on Day 1 of Cohort 3 after the safety review of Cohort 2.
  Interventions: Drug: Tofersen
- Part A-SAD: Cohort 4: Tofersen 60 mg (Experimental): Participants will be administered tofersen 60 mg once by intrathecal bolus injection on Day 1 of Cohort 4 after the safety review of Cohort 3.
  Interventions: Drug: Tofersen
- Part B-MAD: Combined Placebo (Placebo Comparator): Participants will be administered tofersen-matching placebo, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection.
  Interventions: Drug: Placebo
- Part B-MAD: Cohort 5: Tofersen 20 mg (Experimental): Participants will be administered tofersen 20 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection.
  Interventions: Drug: Tofersen
- Part B-MAD: Cohort 6: Tofersen 40 mg (Experimental): Participants will be administered tofersen 40 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety and PK review of Cohort 5.
  Interventions: Drug: Tofersen
- Part B-MAD: Cohort 7: Tofersen 60 mg (Experimental): Participants will be administered tofersen 60 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety, PK review and SOD1 PD review of Cohort 6.
  Interventions: Drug: Tofersen
- Part B-MAD: Cohort 8: Tofersen 100 mg (Experimental): Participants will be administered tofersen 100 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety, PK review and SOD1 PD review of Cohort 7.
  Interventions: Drug: Tofersen
- Part C-Pivotal: Placebo (Placebo Comparator): Participants will be administered tofersen-matching placebo, 3 loading doses administered once every 2 weeks on Days 1, 15, 29 followed by 5 maintenance doses administered once every 4 weeks on Days 57, 85, 113, 141, 169 up to 24 weeks by intrathecal bolus injection.
  Interventions: Drug: Placebo
- Part C-Pivotal: Tofersen 100 mg (Experimental): Participants will be administered tofersen 100 mg, 3 loading doses administered once every 2 weeks on Days 1, 15, 29 followed by 5 maintenance doses administered once every 4 weeks on Days 57, 85, 113, 141, 169 up to 24 weeks by intrathecal bolus injection.
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Administered as specified in the treatment arm.
  Other Names: BIIB067; QALSODY
  Arms: Part A-SAD: Cohort 1: Tofersen 10 mg; Part A-SAD: Cohort 2: Tofersen 20 mg; Part A-SAD: Cohort 3: Tofersen 40 mg; Part A-SAD: Cohort 4: Tofersen 60 mg; Part B-MAD: Cohort 5: Tofersen 20 mg; Part B-MAD: Cohort 6: Tofersen 40 mg; Part B-MAD: Cohort 7: Tofersen 60 mg; Part B-MAD: Cohort 8: Tofersen 100 mg; Part C-Pivotal: Tofersen 100 mg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part A-SAD: Combined Placebo; Part B-MAD: Combined Placebo; Part C-Pivotal: Placebo

SUMMARY:
The primary objectives of Parts A and B of this study are to evaluate the safety, tolerability, and pharmacokinetics (PK) of ascending doses of tofersen in adults with ALS and a documented superoxide dismutase 1 (SOD1) mutation. The primary objective of Part C of this study is to evaluate the clinical efficacy of tofersen administered to adults with ALS and a confirmed SOD1 mutation.

The secondary objective of Parts A and B of this study is to evaluate the effects of tofersen on levels of total SOD1 protein in the cerebrospinal fluid (CSF). The secondary objectives of Part C are to evaluate the safety, tolerability, pharmacodynamic (PD), and biomarker effects of tofersen.

DETAILED DESCRIPTION:
This is a 3-part study to examine the efficacy, safety, tolerability, PK, and PD of tofersen. Part A is the single ascending dose (SAD) component of the study, Part B is the multiple ascending dose (MAD) component of study and Part C is the fixed dose component of the study. Hence, the overall phase of development of the study is 1/2/3.

The study completed on 16 Jul 2021. In total, the study enrolled 176 participants, of which 108 enrolled in Part C.

ELIGIBILITY:
Key Inclusion Criteria: Part A and B

* Weakness attributable to ALS and documented SOD1 mutation at Screening Visit 2.
* A forced vital capacity (FVC) ≥50% of predicted value as adjusted for sex, age, and height (from the sitting position). Participants with stable FVC <50% but ≥45%, whose FVC has not declined by more than 5% in the last 6 months may be considered for inclusion, at the discretion of the Investigator.
* If taking riluzole, participant must be on a stable dose for ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit.
* Medically able to undergo the study procedures, and to adhere to the visit schedule at the time of study entry, as determined by the Investigator.

Key Exclusion Criteria: Part A and B

* History of or positive test result for human immunodeficiency virus.
* History of, or positive test result at Screening, for hepatitis C virus antibody.
* Current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]). Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive hepatitis B surface antibody immunoglobulin G, and positive HBcAb) or vaccination (defined as positive anti-HBs) are eligible to participate in the study.
* Treatment with another investigational drug, biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Specifically, no prior treatment with small interfering ribonucleic acid, stem cell therapy, or gene therapy is allowed.
* Current enrollment in any other interventional study.
* Current or recent (within 1 month) use, or anticipated need, in the opinion of the Investigator, of copper (II) (diacetyl-bis (N4-methylthiosemicarbazone)) or pyrimethamine.
* Current or anticipated need, in the opinion of the Investigator, of a diaphragm pacing system (DPS) during the study period.

Key Inclusion Criteria: Part C

* Weakness attributable to ALS and confirmed SOD1 mutation at Screening Visit.
* If taking riluzole, participant must be on a stable dose for ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit.
* If taking edaravone, participant must have initiated edaravone ≥60 days (2 treatment cycles) prior to Day 1 and expected to remain at that dose until the final study visit, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study. Edaravone may not be administered on dosing days of this study.
* Medically able to undergo the study procedures and to adhere to the visit schedule at the time of study entry, as determined by the Investigator.

Key Exclusion Criteria: Part C

* History of or positive test result for human immunodeficiency virus.
* Current hepatitis C infection (defined as positive hepatitis C virus [HCV] antibody and detectable HCV ribonucleic acid [RNA]). Participants with positive HCV antibody and undetectable HCV RNA are eligible to participate in the study (United States Centers for Disease Control and Prevention).
* Current hepatitis B infection (defined as positive for HBsAg and/or anti-HBc). participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive anti-HBs) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study.
* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use programs), biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Specifically, no prior treatment with small interfering RNA, stem cell therapy, or gene therapy is allowed.
* Current enrollment in any other interventional study.
* Current or recent (within 1 month) use, or anticipated need, in the opinion of the Investigator, of copper (II) (diacetyl-bis(N4-methylthiosemicarbazone)) or pyrimethamine.
* Current or anticipated need, in the opinion of the Investigator, of a DPS during the study period.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (40):
- United States (20):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, P.C., Lincoln, Nebraska
  - Columbia University Medical Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence ALS Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - New Orleans Center for Clinical Research/Volunteer Research Group, an AMR Company, Knoxville, Tennessee
  - Methodist Neurological Institute, Houston, Texas
- Westmead Hospital, Westmead, New South Wales, Australia
- UZ Leuven, Leuven, Belgium
- Canada (4):
  - University of Calgary - Health Sciences Centre, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- Bispebjerg Hospital, Copenhagen, Denmark
- Hopital Pitie Salpetriere, Paris, France
- University of Ulm, Ulm, Baden-Wurttemberg, Germany
- ALS Center - Dept. of Neuroscience "Rita Levi Montalcini", University of Turin, Torino, Italy
- Japan (5):
  - The University of Tokyo Hospital, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kagoshima
  - Research Site, Shinjuku-ku
  - Research Site, Suita-Shi
- Research Site, Warsaw, Poland
- South Korea (2):
  - Research Site, Yangsan, Gyeongsangnam-do
  - Research Site, Seoul
- United Kingdom (2):
  - Research Site, London, Greater London
  - Research Site, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Miller TM, Cudkowicz ME, Shaw PJ, Genge A, Sobue G, Bucelli RC, Chio A, Van Damme P, Ludolph AC, Glass JD, Andrews JA, Babu S, Benatar M, McDermott CJ, Salachas F, Bruneteau G, Al-Chalabi A, Amorin M, Nestorov I, Graham D, Lin L, Sun P, McNeill M, Malek S, Inra J, Garafalo S, Fradette S; VALOR and OLE Working Group. Long-Term Tofersen in SOD1 Amyotrophic Lateral Sclerosis. JAMA Neurol. 2026 Feb 1;83(2):115-125. doi: 10.1001/jamaneurol.2025.4946. PMID 41661214
- [Derived] Miller TM, Cudkowicz ME, Genge A, Shaw PJ, Sobue G, Bucelli RC, Chio A, Van Damme P, Ludolph AC, Glass JD, Andrews JA, Babu S, Benatar M, McDermott CJ, Cochrane T, Chary S, Chew S, Zhu H, Wu F, Nestorov I, Graham D, Sun P, McNeill M, Fanning L, Ferguson TA, Fradette S; VALOR and OLE Working Group. Trial of Antisense Oligonucleotide Tofersen for SOD1 ALS. N Engl J Med. 2022 Sep 22;387(12):1099-1110. doi: 10.1056/NEJMoa2204705. PMID 36129998
- [Derived] Miller T, Cudkowicz M, Shaw PJ, Andersen PM, Atassi N, Bucelli RC, Genge A, Glass J, Ladha S, Ludolph AL, Maragakis NJ, McDermott CJ, Pestronk A, Ravits J, Salachas F, Trudell R, Van Damme P, Zinman L, Bennett CF, Lane R, Sandrock A, Runz H, Graham D, Houshyar H, McCampbell A, Nestorov I, Chang I, McNeill M, Fanning L, Fradette S, Ferguson TA. Phase 1-2 Trial of Antisense Oligonucleotide Tofersen for SOD1 ALS. N Engl J Med. 2020 Jul 9;383(2):109-119. doi: 10.1056/NEJMoa2003715. PMID 32640130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in the Belgium, Canada, Denmark, France, Germany, Italy, Japan, United Kingdom, and the United States from 20 January 2016 to 16 July 2021.
Pre-assignment Details: Study included SAD (Part A), MAD (Part B) and pivotal portions (Part C). Total 176 participants were randomized: 20 into Part A, 50 into Part B including 2 participants who completed Part A, were randomized in Part B after 12-week washout period, hence 2 participants were analysed in both Parts A, B (for total of 68 in Parts A, B), Part C randomized 108 participants.
Groups:
- Part A-SAD: Combined Placebo: Participants were administered BIIB067-matching placebo once by intrathecal bolus injection on Day 1 of Cohorts 1, 2, 3, and 4 respectively.
- Part A-SAD: Cohort 1: BIIB067 10 mg: Participants were administered BIIB067 10 mg once by intrathecal bolus injection on Day 1.
- Part A-SAD: Cohort 2: BIIB067 20 mg: Participants were administered BIIB067 20 mg once by intrathecal bolus injection on Day 1 of Cohort 2 after the safety review of Cohort 1.
- Part A-SAD: Cohort 3: BIIB067 40 mg: Participants were administered BIIB067 40 mg once by intrathecal bolus injection on Day 1 of Cohort 3 after the safety review of Cohort 2.
- Part A-SAD: Cohort 4: BIIB067 60 mg: Participants were administered BIIB067 60 mg once by intrathecal bolus injection on Day 1 of Cohort 4 after the safety review of Cohort 3.
- Part B-MAD: Combined Placebo: Participants were administered BIIB067-matching placebo, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection.
- Part B-MAD: Cohort 5: BIIB067 20 mg: Participants were administered BIIB067 20 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection.
- Part B-MAD: Cohort 6: BIIB067 40 mg: Participants were administered BIIB067 40 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety and pharmacokinetic (PK) review of Cohort 5.
- Part B-MAD: Cohort 7: BIIB067 60 mg: Participants were administered BIIB067 60 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety, PK review and superoxide dismutase 1 (SOD1) pharmacodynamic (PD) review of Cohort 6.
- Part B-MAD: Cohort 8: BIIB067 100 mg: Participants were administered BIIB067 100 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety, PK review and SOD1 PD review of Cohort 7.
- Part C-Pivotal: Placebo: Participants were administered BIIB067-matching placebo, 3 loading doses administered once every 2 weeks on Days 1, 15, 29 followed by 5 maintenance doses administered once every 4 weeks on Days 57, 85, 113, 141, 169 up to 24 weeks by intrathecal bolus injection.
- Part C-Pivotal: BIIB067 100 mg: Participants were administered BIIB067 100 mg, 3 loading doses administered once every 2 weeks on Days 1, 15, 29 followed by 5 maintenance doses administered once every 4 weeks on Days 57, 85, 113, 141, 169 up to 24 weeks by intrathecal bolus injection.
Period: Part A (Up to 63 Days)
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Started | 5 | 3 | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 5 | 2 | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Up to 289 Days)
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Started | 0 (Participants who completed Part A did not enter Part B of the study.) | 0 (Participants who completed Part A did not enter Part B of the study.) | 0 (Participants who completed Part A did not enter Part B of the study.) | 0 (Participants who completed Part A did not enter Part B of the study.) | 0 (Participants who completed Part A did not enter Part B of the study.) | 12 (Started indicates the number of participants who were enrolled into Part B of the study.) | 10 (Started indicates the number of participants who were enrolled into Part B of the study.) | 9 (Started indicates the number of participants who were enrolled into Part B of the study.) | 9 (Started indicates the number of participants who were enrolled into Part B of the study.) | 10 (Started indicates the number of participants who were enrolled into Part B of the study.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 10 | 8 | 9 | 8 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Period: Part C (Up to 236 Days)
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 (Participants who completed Part B did not enter Part C of the study.) | 0 (Participants who completed Part B did not enter Part C of the study.) | 0 (Participants who completed Part B did not enter Part C of the study.) | 0 (Participants who completed Part B did not enter Part C of the study.) | 0 (Participants who completed Part B did not enter Part C of the study.) | 36 (Started indicates the number of participants who were enrolled into Part C of the study.) | 72 (Started indicates the number of participants who were enrolled into Part C of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 64
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Consent Withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) populations for parts A, B, and C included all randomized participants who received at least 1 dose or a part of 1 dose of study treatment (BIIB067 or placebo) in Parts A, B, and C respectively. The demographics data reported for Part B arm groups included only the unique participants who were enrolled directly into Part B of the study.
Groups:
- Part B-MAD: Cohort 6: BIIB067 40 mg: Participants were administered BIIB067 40 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety and PK review of Cohort 5.
- Part B-MAD: Cohort 7: BIIB067 60 mg: Participants were administered BIIB067 60 mg, 3 loading doses once every 2 weeks on Days 1, 15, 29 and 2 maintenance doses once every 4 weeks on Days 57 and 85 by intrathecal injection after the safety, PK review and SOD1 PD review of Cohort 6.
- Total: Total of all reporting groups
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 9 | 8 | 9 | 10 | 36 | 72 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.29) | 50.3 (7.64) | 55.3 (17.62) | 49.0 (3.61) | 45.0 (12.82) | 49.2 (11.04) | 42.1 (11.19) | 57.5 (11.75) | 45.6 (10.71) | 48.9 (10.80) | 51.2 (11.57) | 48.1 (12.64) | 49.2 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 1 | 4 | 5 | 3 | 5 | 3 | 6 | 17 | 29 | 78
  Male | 3 | 0 | 3 | 2 | 2 | 7 | 6 | 3 | 6 | 4 | 19 | 43 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5
  Not Hispanic or Latino | 4 | 3 | 3 | 1 | 5 | 9 | 4 | 5 | 4 | 7 | 28 | 47 | 120
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 5 | 3 | 7 | 21 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not reported indicates that race data was not reported due to confidentiality regulations.
  Participants
    Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 5 | 10
    Race: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Race: White | 4 | 3 | 3 | 1 | 5 | 7 | 4 | 4 | 4 | 7 | 25 | 44 | 111
    Race: Not Reported | 1 | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 5 | 3 | 7 | 21 | 51
    Race: Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) [Mean (Standard Deviation); unit: score on a scale] — ALSFRS-R measures respiratory, bulbar function, gross, and fine motor skills. 12 questions, each scored from 0-4 (no-full function), for a total score of 48. Scores decline with disease progression. Higher scores represent better function. Population: Modified ITT (mITT) population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment. This measure was only analyzed for Part C arms groups.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 39 | 60
    (all) |  |  |  |  |  |  |  |  |  |  | 35.4 (5.66) | 36.0 (6.40) | 35.78 (6.109)
Cerebrospinal Fluid (CSF) Levels of Total SOD1 Protein Concentration [Geometric Mean (Full Range); unit: nanograms per milliliter (ng/mL)] — Population: Pharmacodynamic (PD) population is subset of ITT population with at least 1 post-dose PD measurement in Part B. mITT population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment. This measure was only analyzed for Part B and C arms groups.
  nanograms per milliliter (ng/mL)
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 9 | 1 | 1 | 4 | 21 | 39 | 79
    (all) |  |  |  |  |  | 70.40 [57.2 to 87.9] | 102.00 [102.00 to 102.00] | 125.00 [125.00 to 125.00] | 82.80 [82.8 to 82.8] | 135.86 [92.5 to 199.0] | 107.07 [60.0 to 322.0] | 103.32 [38.8 to 282.0] | 104.64 [38.8 to 322.0]
Percentage Predicted Slow Vital Capacity (SVC) [Mean (Standard Deviation); unit: percent predicted] — Population: mITT population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment. This measure was only analyzed for Part C arms groups.
  percent predicted
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 39 | 60
    (all) |  |  |  |  |  |  |  |  |  |  | 83.7 (17.87) | 80.3 (14.22) | 81.50 (15.533)
Handheld Dynamometry (HHD) Megascore as Measured by the HHD Device [Mean (Standard Deviation); unit: score on a scale] — 16 muscle groups were evaluated in upper, lower extremities. Muscle strength values were normalized to Z scores as (post-baseline measurements - mean)/standard deviation (SD), averaged to provide HHD overall megascore. Population: mITT population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment. This measure was only analyzed for Part C arms groups.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 39 | 60
    (all) |  |  |  |  |  |  |  |  |  |  | 0.0 (0.60) | 0.0 (0.67) | -0.007 (0.6396)
Neurofilament Light Chain (NfL) Concentration in Plasma [Geometric Mean (Full Range); unit: picograms per mL (pg/mL)] — Population: mITT population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment. This measure was only analyzed for Part C arms groups.
  picograms per mL (pg/mL)
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 39 | 60
    (all) |  |  |  |  |  |  |  |  |  |  | 92.7 [9 to 370] | 121.8 [12 to 329] | 110.49 [8.8 to 370.4]

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE is any untoward medical occurrence that at any dose results in death, life-threatening event, requires inpatient hospitalization, significant disability/incapacity or congenital anomaly.
Time Frame: Part A: First dose up to Day 63; Part B: First dose up to Day 289
Population: Safety population included all randomized participants who received at least 1 dose or a part of 1 dose of study treatment (BIIB067 or placebo) in Part A or B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants
  AEs | 2 | 2 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
  SAEs | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0

2. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinical laboratory assessments included hematology, chemistry, and urinalysis.
Time Frame: Part A: Up to Day 57; Part B: Up to Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants
  Pleocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Eosinophilia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood Phosphorus Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CSF Protein Increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1
  CSF White Blood Cell Count Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
  CSF White Blood Cell Count Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Gamma-Glutamyltransferase Increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine Output Decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: The criteria for clinically significant vital sign abnormalities include: Temperature: >38 degree Celsius (°C) or an increase from baseline of ≥1°C; Pulse: >120 beats per minute (bpm) or an increase from baseline of >20 bpm, <50 bpm or a decrease from baseline of >20 bpm; Systolic blood pressure (BP): >180 mmHg or an increase from baseline of >40 mmHg, <90 mmHg or a decrease from baseline of >30 mmHg; Diastolic BP: >105 mmHg or an increase from baseline of >30 mmHg, <50 mmHg or a decrease from baseline of >20 mmHg.
Time Frame: Part A: Up to Day 57; Part B: Up to Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Clinically significant physical examination abnormalities included weight decreased.
Time Frame: Part A: Up to Day 57; Part B: Up to Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

5. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Neurological Examination Abnormalities
Description: Clinically significant neurological examination abnormalities included hyporeflexia.
Time Frame: Part A: Up to Day 57; Part B: Up to Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant 12-lead Electrocardiograms (ECGs) Abnormalities
Time Frame: Part A: Up to Day 57; Part B: Up to Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 12 | 10 | 9 | 9 | 10
Participants
  Maximum Increase From Baseline QTcF > 30 to 60 ms | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 3
  Maximum Post-baseline QTcF > 480 to 500 ms | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Maximum Observed Concentration (Cmax)
Time Frame: Part A: Pre-dose, 1, 2, 4, 6 hrs post-dose on Day 1; Part B: Pre-dose, 1, 2, 4, 6 hrs post-dose on Day 1 and 1, 2, 4, 6 hrs post-dose on Day 85
Population: PK population is the subset of the ITT population (all randomized participants who received at least 1 dose or a part of 1 dose of study treatment) of participants with at least 1 post-dose PK measurement in Part A or B. Data was not collected for participants on Day 85 for Part A of the study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
ng/mL
  Day 1 | 64.94 [38.8 to 159.0] | 75.06 [43.0 to 144.0] | 202.09 [174.0 to 236.0] | 529.63 [148.0 to 1450.0] | 80.75 [20.1 to 393.0] | 229.41 [26.3 to 948.0] | 437.28 [128.0 to 1930.0] | 1031.74 [285.0 to 3530.0]
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 9 | 10
  Day 85 |  |  |  |  | 112.74 [29.7 to 203.0] | 199.69 [93.6 to 537.0] | 411.00 [74.1 to 1450.0] | 1181.83 [170.0 to 3990.0]

8. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Time to Reach Maximum Observed Concentration (Tmax)
Time Frame: as for outcome 7
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B. Data was not collected for participants on Day 85 for Part A of the study.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hours
  Day 1 | 4.58 [4.0 to 6.0] | 4.16 [2.0 to 6.0] | 6.00 [6.0 to 6.0] | 2.70 [2.0 to 6.0] | 7.01 [2.0 to 24.0] | 3.68 [1.0 to 6.0] | 2.44 [1.0 to 6.0] | 3.67 [1.0 to 24.0]
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 9 | 10
  Day 85 |  |  |  |  | 3.93 [2.0 to 6.0] | 3.97 [1.0 to 6.0] | 3.12 [1.0 to 6.0] | 3.82 [1.0 to 6.0]

9. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Area Under the Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h)
Time Frame: Parts A and B: Pre-dose, 1, 2, 4, 6 hrs post-dose on Day 1
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B.
Measure: Geometric Mean (Full Range); unit: hour*ng/mL
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hour*ng/mL | 879.86 [550.8 to 1989.5] | 1027.18 [879.2 to 1263.2] | 2873.77 [2347.2 to 3543.4] | 5196.11 [2410.2 to 10977.3] | 1009.85 [372.8 to 2192.3] | 2875.13 [541.1 to 6984.8] | 4289.16 [1347.6 to 10637.1] | 11344.47 [4025.5 to 26143.0]

10. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Time Frame: Part A: Pre-dose Day 1, Days 29 and 57; Part B: Pre-dose Days 1, 15, 29, 57 and 85; Day 106 and 169
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hour*ng/mL | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values. | NA (NA) — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the AUC0-infinity values.

11. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast)
Time Frame: Part A: Pre-dose Day 1, Days 29 and 57; Part B: Pre-dose Days 1, 15, 29, 57 and 85; Day 106 and 169
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hour*ng/mL | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful. | NA (NA) — Due to the large number of values below the level of quantification at various times, the last measurable concentration would have varied across individuals which makes this parameter not useful.

12. Primary Outcome: Parts A and B: PK Parameter of BIIB067 in Plasma: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: Part A: Pre-dose Day 1, Days 29 and 57; Part B: Pre-dose Days 1, 15, 29, 57 and 85; Day 106 and 169
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hours | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the apparent terminal t1/2 values.

13. Primary Outcome: Parts A and B: PK Parameters of BIIB067 in CSF Levels: Terminal Elimination Half-life (t1/2)
Time Frame: Part A: Pre-dose Day 1, Days 29 and 57; Part B: Pre-dose Days 1, 15, 29, 57 and 85; Day 106 and 169
Population: PK population is the subset of the ITT population with at least 1 post-dose PK measurement in Part A or B.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 10 | 9 | 9 | 10
hours | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values. | NA [NA to NA] — Data is not available as the concentration values were below the level of quantification and could not be quantified to estimate the terminal t1/2 values.

14. Primary Outcome: Part C: Change From Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Total Score at Week 28
Description: The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are 12 questions, each scored from 0 (no function) to 4 (full function), for a total possible score of 48. Scores decline with disease progression. ALSFRS-R scores calculated at diagnosis can be compared to scores throughout time to determine the speed of progression. Higher scores represent better function, negative change from baseline indicates disease progression.
Time Frame: Baseline, Week 28 (Day 197)
Population: mITT population included all participants who met the prognostic enrichment criteria for rapid disease progression in Part C who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
score on scale | -8.1 (1.79) | -7.0 (1.42)
Statistical Analysis 1: Comparison: Part C-Pivotal: Placebo vs Part C-Pivotal: BIIB067 100 mg; Joint rank test combining function and mortality were used for statistical inference and the estimates were from the Analysis of covariance (ANCOVA) for change from baseline. Multiple imputation was used to handle missing data for withdrawals other than death in the joint rank analysis. Multiple imputation was used to handle all missing data in the ANCOVA for change from baseline; Test type: Superiority; p = 0.9689, Joint rank — Joint rank p-value was calculated from ANCOVA model which included treatment as fixed effect, adjusts for covariates: Baseline disease duration since symptom onset, baseline ALSFRS-R total score, and use of riluzole or edaravone; least square (LS) mean difference = 1.2, 95% CI 2-sided [-3.19 to 5.53], Standard Error of Mean 2.22 — ANCOVA model included treatment as a fixed effect, adjusts for the covariates: Baseline disease duration since symptom onset, baseline ALSFRS-R total score, and use of riluzole or edaravone

15. Secondary Outcome: Part B: CSF Levels of Total SOD1 Protein Concentration Ratio to Baseline
Description: Total CSF SOD1 protein ratio to baseline was calculated.
Time Frame: Day 85
Population: PD population is the subset of the ITT population with at least 1 post-dose PD measurement in Part B.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg
Number analyzed (Participants) | 12 | 10 | 9 | 8 | 10
ratio | 0.97 [0.83 to 1.13] | 0.99 [0.83 to 1.18] | 0.73 [0.61 to 0.87] | 0.79 [0.66 to 0.94] | 0.64 [0.55 to 0.76]
Statistical Analysis 1: Comparison: Part B-MAD: Combined Placebo vs Part B-MAD: Cohort 5: BIIB067 20 mg; Difference in LS geometric mean ratio (BIIB067:Placebo) was calculated; Test type: Superiority; p < 0.0001, Wilcoxon rank sum test; Difference in LS geometric mean ratio = 0.67, 95% CI 2-sided [0.53 to 0.84]
Statistical Analysis 2: Comparison: Part B-MAD: Combined Placebo vs Part B-MAD: Cohort 6: BIIB067 40 mg; Difference in LS geometric mean ratio (BIIB067:Placebo) was calculated; Test type: Superiority; p = 0.0002, Wilcoxon rank sum test; Difference in LS geometric mean ratio = 0.75, 95% CI 2-sided [0.60 to 0.95]
Statistical Analysis 3: Comparison: Part B-MAD: Combined Placebo vs Part B-MAD: Cohort 7: BIIB067 60 mg; Difference in LS geometric mean ratio (BIIB067:Placebo) was calculated; Test type: Superiority; p = 0.0641, Wilcoxon rank sum test; Difference in LS geometric mean ratio = 0.81, 95% CI 2-sided [0.65 to 1.02]
Statistical Analysis 4: Comparison: Part B-MAD: Combined Placebo vs Part B-MAD: Cohort 8: BIIB067 100 mg; Difference in LS geometric mean ratio (BIIB067:Placebo) was calculated; Test type: Superiority; p < 0.0001, Wilcoxon rank sum test; Difference in LS geometric mean ratio = 0.67, 95% CI 2-sided [0.53 to 0.84]

16. Secondary Outcome: Part C: CSF Levels of Total SOD1 Protein Concentration Ratio to Baseline
Description: Total CSF SOD1 protein ratio to baseline was calculated and LS Geometric Mean ratio to baseline was reported.
Time Frame: Week 28 (Day 197)
Population: as for outcome 14
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
ratio | 1.16 [0.96 to 1.40] | 0.71 [0.62 to 0.83]
Statistical Analysis 1: Comparison: Part C-Pivotal: Placebo vs Part C-Pivotal: BIIB067 100 mg; The ANCOVA model included covariates for the corresponding baseline value i.e. log value, baseline disease duration since symptom onset, and use of riluzole or edaravone. Multiple imputation was used to handle missing data for withdrawals. Difference in LS geometric mean ratio to baseline (BIIB067:Placebo) was calculated; Test type: Superiority; p < 0.0001, ANCOVA — The analysis was based on ANCOVA model with natural log transformed data. P-value for this secondary outcome measure (OM) is nominal as statistical significance was not met on the primary OM; Difference in LS geometric mean ratio = 0.62, 95% CI 2-sided [0.49 to 0.78]

17. Secondary Outcome: Part C: Neurofilament Light Chain (NfL) Plasma Concentration Ratio to Baseline
Description: NfL is a biomarker whose concentration was assessed in plasma. Plasma NfL ratio to baseline was calculated.
Time Frame: Baseline, Day 197 (Week 28)
Population: as for outcome 14
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
ratio | 1.20 [0.94 to 1.52] | 0.40 [0.33 to 0.48]
Statistical Analysis 1: Comparison: Part C-Pivotal: Placebo vs Part C-Pivotal: BIIB067 100 mg; Difference in LS geometric mean ratio (BIIB067:Placebo) was calculated; Test type: Superiority; p < 0.0001, ANCOVA — The analysis was based on ANCOVA model with natural log transformed data. The model included covariates for the corresponding baseline value i.e. log value, baseline disease duration since symptom onset, and use of riluzole or edaravone; P-value for this secondary OM is nominal as statistical significance was not met on the primary OM; Difference in LS geometric mean ratio = 0.33, 95% CI 2-sided [0.25 to 0.45]

18. Secondary Outcome: Part C: Change From Baseline in Percent Predicted Slow Vital Capacity (SVC) at Week 28
Description: Vital capacity was measured by means of an SVC test, administered in the upright position.
Time Frame: Baseline, Week 28 (Day 197)
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
percent predicted | -22.20 (4.771) | -14.31 (3.557)
Statistical Analysis 1: Comparison: Part C-Pivotal: Placebo vs Part C-Pivotal: BIIB067 100 mg; Joint rank test combining function and mortality were used for statistical inference and the estimates were from the ANCOVA for change from baseline. Multiple imputation was used to handle missing data for withdrawals other than death in the joint rank analysis. Multiple imputation was used to handle all missing data in the ANCOVA for change from baseline; Test type: Superiority; p = 0.3233, Joint rank — Joint rank p-value was calculated from ANCOVA model which included treatment as fixed effect, adjusts for covariates: Baseline disease duration since symptom onset, baseline ALSFRS-R total score, baseline SVC, and use of riluzole or edaravone; P-value for this secondary OM is nominal as statistical significance was not met on the primary OM; LS mean difference = 7.90, 95% CI 2-sided [-3.528 to 19.322], Standard Error of Mean 5.829 — ANCOVA model included treatment as a fixed effect, adjusts for the covariates: Baseline disease duration since symptom onset, baseline ALSFRS-R total score, baseline SVC, and use of riluzole or edaravone

19. Secondary Outcome: Part C: Change From Baseline in Handheld Dynamometry (HHD) Megascore as Measured by the HHD Device at Week 28
Description: Quantitative muscle strength was evaluated using HHD, which tests isometric strength of multiple muscles using standard participant positioning. Sixteen muscle groups were evaluated in both upper and lower extremities. The muscle strength values were normalized to Z scores as (post-baseline measurements - mean)/SD and averaged to provide HHD overall megascore. The overall megascore was created by averaging all eight bilateral measurement Z scores, if no more than 10 (≤ 10) measures are missing. A negative change from baseline indicated decreased muscle strength.
Time Frame: Baseline, Week 28 (Day 197)
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
score on a scale | -0.37 (0.096) | -0.34 (0.073)
Statistical Analysis 1: Comparison: Part C-Pivotal: Placebo vs Part C-Pivotal: BIIB067 100 mg; Test type: Superiority; p = 0.8390, ANCOVA — ANCOVA model included treatment as fixed effect and adjusts for following covariates: Baseline disease duration since symptom onset, baseline HHD overall megascore, and use of riluzole/edaravone. Missing data were handled using multiple imputation; P-value for this secondary OM is nominal as statistical significance was not met on the primary OM; LS mean difference = 0.02, 95% CI 2-sided [-0.207 to 0.255], Standard Error of Mean 0.118

20. Secondary Outcome: Part C: Time to Death or Permanent Ventilation
Description: Time to Death or Permanent Ventilation is defined as the time to the earliest occurrence of one of the following events that were adjudicated by an independent committee: Death; Permanent ventilation (≥22 hours of mechanical ventilation [invasive or noninvasive] per day for ≥21 consecutive days).
Time Frame: Baseline up to Week 28 (Day 197)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
days | NA [NA to NA] — Not estimated due to insufficient number of participants with events. | NA [NA to NA] — Not estimated due to insufficient number of participants with events.

21. Secondary Outcome: Part C: Time to Death
Time Frame: Baseline up to Week 28 (Day 197)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 21 | 39
days | NA [NA to NA] — Not estimated due to insufficient number of participants with events. | NA [NA to NA] — Not estimated due to insufficient number of participants with events.

22. Secondary Outcome: Part C: Number of Participants Experiencing AEs and SAEs
Description: as for outcome 1
Time Frame: First dose up to Day 236
Population: Safety population included all participants in Part C who were randomized and received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
Participants
  AEs | 34 | 69
  SAEs | 5 | 13

ADVERSE EVENTS:
Time Frame: Part A: First dose up to Day 63; Part B: First dose up to Day 289; Part C: First dose up to Day 236
Description: Safety population included all randomized participants who received at least 1 dose or a part of 1 dose of study treatment (BIIB067 or placebo) in Part A or B. Safety population included all participants in Part C who were randomized and received at least one dose of study treatment. MedDRA version for Parts A and B: 22.0, Part C: 24.0
Arm/Group | Part A-SAD: Combined Placebo | Part A-SAD: Cohort 1: BIIB067 10 mg | Part A-SAD: Cohort 2: BIIB067 20 mg | Part A-SAD: Cohort 3: BIIB067 40 mg | Part A-SAD: Cohort 4: BIIB067 60 mg | Part B-MAD: Combined Placebo | Part B-MAD: Cohort 5: BIIB067 20 mg | Part B-MAD: Cohort 6: BIIB067 40 mg | Part B-MAD: Cohort 7: BIIB067 60 mg | Part B-MAD: Cohort 8: BIIB067 100 mg | Part C-Pivotal: Placebo | Part C-Pivotal: BIIB067 100 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 0/3 | 0/6 | 1/12 | 1/10 | 0/9 | 1/9 | 0/10 | 0/36 | 1/72
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 0/3 | 0/6 | 2/12 | 2/10 | 1/9 | 2/9 | 0/10 | 5/36 | 13/72
Other Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 3/3 | 3/3 | 6/6 | 11/12 | 10/10 | 9/9 | 9/9 | 10/10 | 34/36 | 68/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-SAD: Combined Placebo (N=5) | Part A-SAD: Cohort 1: BIIB067 10 mg (N=3) | Part A-SAD: Cohort 2: BIIB067 20 mg (N=3) | Part A-SAD: Cohort 3: BIIB067 40 mg (N=3) | Part A-SAD: Cohort 4: BIIB067 60 mg (N=6) | Part B-MAD: Combined Placebo (N=12) | Part B-MAD: Cohort 5: BIIB067 20 mg (N=10) | Part B-MAD: Cohort 6: BIIB067 40 mg (N=9) | Part B-MAD: Cohort 7: BIIB067 60 mg (N=9) | Part B-MAD: Cohort 8: BIIB067 100 mg (N=10) | Part C-Pivotal: Placebo (N=36) | Part C-Pivotal: BIIB067 100 mg (N=72)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired self-care (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis chemical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Csf protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Csf white blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-SAD: Combined Placebo (N=5) | Part A-SAD: Cohort 1: BIIB067 10 mg (N=3) | Part A-SAD: Cohort 2: BIIB067 20 mg (N=3) | Part A-SAD: Cohort 3: BIIB067 40 mg (N=3) | Part A-SAD: Cohort 4: BIIB067 60 mg (N=6) | Part B-MAD: Combined Placebo (N=12) | Part B-MAD: Cohort 5: BIIB067 20 mg (N=10) | Part B-MAD: Cohort 6: BIIB067 40 mg (N=9) | Part B-MAD: Cohort 7: BIIB067 60 mg (N=9) | Part B-MAD: Cohort 8: BIIB067 100 mg (N=10) | Part C-Pivotal: Placebo (N=36) | Part C-Pivotal: BIIB067 100 mg (N=72)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 6 | 9
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 2 | 12
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Dust allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Gastric infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 7 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Systemic viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 2 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 5 | 15 | 17
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 11 | 13
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 3
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 3 | 5 | 4 | 1 | 4 | 7 | 21 | 41
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Csf protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 6
Csf white blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 7
Csf white blood cell count positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 5 | 2 | 15
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 3 | 6 | 19
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 4
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 7 | 4 | 2 | 4 | 6 | 16 | 33
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleocytosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 4
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 2
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT02623699/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT02623699/SAP_001.pdf